CLINICAL TRIAL: NCT03207919
Title: The Lullaby Project: A Musical Intervention for Pregnant Women
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Virginia Commonwealth University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: HM20008253
Record Dates: First submitted 2017-06-29; First posted 2017-07-05 (Actual); Last update posted 2018-04-24 (Actual); Status verified 2018-04

CONDITIONS: Pregnancy Related
Keywords: maternal-fetal attachment; maternal health; maternal stress; Lullaby Project

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Lullaby Project (Experimental)
  Interventions: Behavioral: Lullaby Project
- Control Group (No Intervention)

INTERVENTIONS:
Behavioral: Lullaby Project — Pregnant women will participate in 3 group sessions. They will write and record a lullaby, and then listen to each recorded lullaby and reflect on their experience.
  Arms: Lullaby Project

SUMMARY:
This study will evaluate the potential impact of a brief musical intervention, the Lullaby Project, in a sample of pregnant women. The study aims are:

1. To determine the potential effect of the Lullaby Project on maternal-fetal attachment.
2. To evaluate the potential impact of the Lullaby Project on maternal mental health.
3. To characterize the potential impact of the Lullaby Project on perceived maternal stress.

DETAILED DESCRIPTION:
Music has the power to build a sense of community and belonging - a crucial process in a U.S. that is steadily becoming more diverse. In America, there is no more pressing issue for children's development than their families' access to basic needs: housing, food, safety and health, as well as education. While music may seem a long way from living wages or immigration reform, the arts, including music, have a substantial role to play in building healthy families.

Over the last three years, musicians from Carnegie Hall's Weill Music Institute have developed the Lullaby Project, in which mothers living in challenging circumstances have the opportunity to write and record a song for their babies or very young children. As of spring 2015, more than 150 lullabies have been created in hospitals, correctional facilities, shelters, programs for teen parents, and other settings where young families face challenges every day. The purpose of this music-based intervention is to initiate or encourage and support the bonding process, to support parents' aspirations to create the family they want for their children, and to harness their creativity as a tool for imagining and building future possibilities.

This study proposes an arts-based intervention to improve maternal-child attachment. Based on theory from the arts and evidence from psychology and pediatrics, this intervention will test the ability of music creation to stimulate maternal attitudes regarding parenting, scores for attachment, and symptoms of anxiety, depression, and stress. In addition, the intervention will focus on at-risk women and their families with a goal of providing a healthier start for their children and preventing transition of these parents and children into the high-risk group.

Patients who consent to participate will be randomly assigned in a 1:1 ratio to participate in an intervention or control group. Each participant will be asked to complete a self-report battery of questionnaires pertaining to their pregnancy, mental health, and perceived stress. At the completion of the questionnaires, referral information for mental health support will be provided to all participants.

Women randomized to the intervention will participate in the three group sessions described below with approximately 8-10 other pregnant women at Virginia Commonwealth University.

i. Session 1: (5 hours) Participants collaborate with project musicians to compose an original lullaby. Efforts will be made to have a 1:1 musician-participant ratio, however, depending on group size, two participants may be paired with one musician.

ii. Session 2: (5 hours) Participants collaborate with project musicians to refine and record their lullaby. The recorded lullaby will not be collecting as data, nor will it be stored as such for this study. No other recordings will be made during the course of this study.

iii. Session 3: (2 hours) Participants listen to each recorded lullaby and are invited to informally reflect on their experience, both individually with one research staff member (study or project coordinator), and within the group.

ELIGIBILITY:
Inclusion Criteria:

* Age: at least 18 years of age.
* Must be able to read and understand English, and provide informed consent.
* Must be in the second or third trimester of pregnancy.

Exclusion Criteria:

* Age: Under the age of 18.
* Unable to read and understand English, and provide informed consent.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 44 (Actual)
Dates: Start 2016-11-04 (Actual); Primary Completion 2017-05-15 (Actual); Study Completion 2017-05-15 (Actual)

PRIMARY OUTCOMES:
Maternal Fetal Attachment | End of Study (2 months)
  As assessed by the Maternal Fetal Attachment Scale (MFAS)

SECONDARY OUTCOMES:
Mental Health | End of Study (2 months)
  General psychiatric distress as assessed by the Symptom Checklist (SCL-27)
Perceived Maternal Stress | End of Study (2 months)
  As assessed by the Perceived Stress Scale (PSS)

CONTACTS AND LOCATIONS:
Overall Officials: Jennifer L Hinesley, Psy. D, Principal Investigator — Virginia Commonwealth University
Locations (1):
- Virginia Commonwealth University, Richmond, Virginia, United States